CLINICAL TRIAL: NCT01227707
Title: An Open-label Study to Assess the Effect of Combination Treatment With Avastin and Xeloda, Plus Pre-operative Standard Radiotherapy, on Response Rate in Patients With Locally Advanced Rectal Cancer.
Brief Title: A Study of Avastin (Bevacizumab) Plus Xeloda (Capecitabine) in Patients With Locally Advanced Rectal Cancer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML18522
Record Dates: First submitted 2010-10-22; First posted 2010-10-25 (Estimated); Results first posted 2014-08-15 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-07

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Capecitabine; Radiotherapy; Fluorouracil; Leucovorin

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: bevacizumab [Avastin]; Drug: capecitabine [Xeloda]; Radiation: Radiation therapy; Procedure: Mesorectal excision; Drug: 5-fluorouracil; Drug: leucovorin

INTERVENTIONS:
Drug: bevacizumab [Avastin] — 5 mg/kg intravenously every 2 weeks, 4 cycles
Drug: capecitabine [Xeloda] — 825 mg/m2 twice daily orally, 38 days
Radiation: Radiation therapy — Total dose of 45 Gy over 38 days
Procedure: Mesorectal excision — 6-8 weeks after completion of neoadjuvant treatment
Drug: bevacizumab [Avastin] — Post-surgery adjuvant treatment at the discretion of the investigator: 5 mg/kg iv every 2 weeks for at least 6 months
Drug: 5-fluorouracil — Post-surgery adjuvant therapy: bolus of 400mg/m2 iv plus iv infusion of 600 mg/m2 on Days 1 and 2 of each 2-week cycle for 6 months
Drug: leucovorin — Post-surgery adjuvant treatment: 100 mg/m2 iv on Days 1 and 2 of each 2-week cycle for 6 months

SUMMARY:
This open-label study will assess the efficacy and safety of Avastin (bevacizumab) plus Xeloda (capecitabine) in combination with standard technique radiotherapy of the pelvic region in the neo-adjuvant setting in patients with locally advanced primary rectal cancer. Patients will receive 4 courses of Avastin at a dose of 5 mg/kg intravenously (iv) every 2 weeks and for 38 days Xeloda at dose of 825 mg/kg twice daily orally, plus radiation therapy. After surgery, adjuvant treatment with 5-fluorouracil/leucovorin and, at the discretion of the investigator, with Avastin 5 mg/kg iv every 2 weeks for at least 6 months will be given.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >=18 years of age
* Patients with confirmed rectal cancer who are subject to surgery and would benefit from pre-operative combined chemo-radiotherapy
* Measurable and/or evaluable lesions according to RECIST criteria
* EOCG performance status 0-1

Exclusion Criteria:

* Prior radiotherapy or chemotherapy for rectal cancer
* Untreated brain metastases or spinal cord compression or primary brain tumors
* Chronic daily treatment with high-dose aspirin (>325 mg/day) or other medications known to predispose to gastrointestinal ulceration
* Co-existing malignancies, or malignancies diagnosed within the last 5 years, with the exception of basal and squamous cell cancer, or cervical cancer in situ.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2005-11; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (9):
- Italy (9):
  - Ancona
  - Bologna
  - Cuneo
  - Genova
  - Napoli
  - Paola
  - Pisa
  - Roma
  - Siena

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab (Bv)+Capecitabine/Bv+Leucovorin+5-fluorouracil: Participants received bevacizumab 5 milligrams per kilogram (mg/kg) intravenously (IV) on Days -14, 1, 15, and 29 and capecitabine 825 milligrams per square meter (mg/m^2) orally (PO) twice daily (BID) from Days 1 to 38. Participants also received radiation therapy given at a daily fraction of 1.8 Gray (Gy) administered in 5 weekly fractions starting at Week 1 (through Week 6) for a maximum total dose of 45 Gy. Six to 8 weeks following all above treatments, participants received complete mesorectal excision surgery. After surgery, participants received bevacizumab 5 mg/kg IV on Day 1 and leucovorin 100 mg/m^2 IV (over 2 hours) followed by 5-fluorouracil (5-FU) 400 mg/m^2 IV bolus and then 5-FU 600 mg/m^2 IV (over 22 hours) on Days 1 and 2 every 2 weeks for a maximum of 12 cycles.
Period: Overall Study
Arm/Group | Bevacizumab (Bv)+Capecitabine/Bv+Leucovorin+5-fluorouracil
Started | 43
Completed | 19
Not Completed | 24
Not completed — Adverse Event | 10
Not completed — Progression of disease | 3
Not completed — Withdrawal by Subject | 1
Not completed — Patient non-compliance | 3
Not completed — Medical decision | 6
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) population: all participants who were included in the trial by signing the informed consent and were assigned to a study patient number.
Groups:
- Bv+Capecitabine/Bv+Leucovorin+5-FU: Participants received bevacizumab 5 mg/kg IV on Days -14, 1, 15, and 29 and capecitabine 825 mg/m^2 PO BID from Days 1 to 38. Participants also received radiation therapy given at a daily fraction of 1.8 Gy administered in 5 weekly fractions starting at Week 1 (through Week 6) for a maximum total dose of 45 Gy. Six to 8 weeks following all above treatments, participants received complete mesorectal excision surgery. After surgery, participants received bevacizumab 5 mg/kg IV on Day 1 and leucovorin 100 mg/m^2 IV (over 2 hours) followed by 5-FU 400 mg/m^2 IV bolus and then 5-FU 600 mg/m^2 IV (over 22 hours) on Days 1 and 2 every 2 weeks for a maximum of 12 cycles.
Arm/Group | Bv+Capecitabine/Bv+Leucovorin+5-FU
Number analyzed (Participants) | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.49 (10.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 25

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Pathological Complete Response (pCR)
Description: pCR was defined as the absence of viable tumor cells, as determined by standard histologic procedure, in the tumor specimen (including regional lymph nodes) obtained at surgery. In order to minimize evaluation bias, tumor specimens were analyzed by both a central and local pathologist. The number of participants with pathological tumor stage 0 (pT0) and regional lymph nodes stage 0 (pN0) at surgery was determined. pCR was defined as the number of participants with pT0 and pN0 at surgery divided by the total number of participants with pathological tumor stage data collected.
Time Frame: 6 to 8 weeks following completion of neoadjuvant treatment
Population: ITT population; only participants who underwent surgery and had pathological tumor stage data were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bv+Capecitabine/Bv+Leucovorin+5-FU
Number analyzed (Participants) | 40
percentage of participants | 10.00 [2.79 to 23.66]
Statistical Analysis 1: Comparison: Bv+Capecitabine/Bv+Leucovorin+5-FU; Test type: Superiority or Other; p = 1.00, one sample binomial test

2. Secondary Outcome: Percentage of Participants by Primary Tumor (T), Regional Lymph Nodes (N), and Distant Metastasis (M) Clinical Stage at Baseline and at the End of Neo-Adjuvant Treatment (NAT)
Description: The frequencies of clinical tumor stage T (0, 1, 2, 3, 4, or X), regional lymph nodes stage N (0, 1, 2, 3, or 4), and distant metastasis clinical stage M (0, 1, or X) at baseline and at the end of NAT were assessed. The frequencies of pathological tumor stage T and regional lymph nodes stage N at surgery were evaluated. The clinical tumor and lymph node status was assessed by clinical examination, endosonography, and/or rectosigmoidoscopy, and pelvic and abdomen computerized tomography (CT) scan or magnetic resonance imaging (MRI). Response to treatment had to be assessed within 6 weeks after end of treatment by using the same techniques performed at baseline.
Time Frame: Baseline (BL) and end of neoadjuvant treatment (within 6 weeks after the completion of study treatment)
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Bv+Capecitabine/Bv+Leucovorin+5-FU
Number analyzed (Participants) | 43
percentage of participants
  Baseline: T0, N0 | 0
  End of NAT: T0, N0 | 4.65
  Baseline: T1, N0 | 0
  End of NAT: T1, N0 | 4.65
  Baseline: T1, NX | 0
  End of NAT: T1, NX | 2.33
  Baseline: T2, N0 | 0
  End of NAT: T2, N0 | 18.60
  Baseline: T2, N1 | 9.30
  End of NAT: T2, N1 | 9.30
  Baseline: T2, NX | 0
  End of NAT: T2, NX | 6.98
  Baseline: T3, N0 | 32.56
  End of NAT: T3, N0 | 18.60
  Baseline: T3, N1 | 46.51
  End of NAT: T3, N1 | 9.30
  Baseline: T3, N2 | 0
  End of NAT: T3, N2 | 2.33
  Baseline: T3, NX | 2.33
  End of NAT: T3, NX | 6.98
  Baseline: T4, N0 | 0
  End of NAT: T4, N0 | 4.65
  Baseline: T4, N1 | 2.33
  End of NAT: T4, N1 | 0
  Baseline: T4, N2 | 2.33
  End of NAT: T4, N2 | 0
  Baseline: T4, N3 | 2.33
  End of NAT: T4, N3 | 0
  Baseline: TX, N0 | 0
  End of NAT: TX, N0 | 2.33
  Baseline: TX, N2 | 2.33
  End of NAT: TX, N2 | 0
  Baseline: M0 | 97.67
  End of NAT: M0 | 81.40
  Baseline: M1 | 2.33
  End of NAT: M1 | 2.33
  Baseline: MX | 0
  End of NAT: MX | 9.30

3. Secondary Outcome: Percentage of Participants Undergoing Sphincter-Saving Surgery by Type of Procedure
Time Frame: 6 to 8 weeks after completion of study treatment
Population: ITT population; only participants who underwent surgery were included in the analysis. n (number) equals (=) number of participants assessed for the specified parameter (colostomy)
Measure: Number; unit: percentage of participants
Arm/Group | Bv+Capecitabine/Bv+Leucovorin+5-FU
Number analyzed (Participants) | 40
percentage of participants
  Anterior resection | 70.0
  Abdomen-peritoneal amputation (Miles) | 22.5
  Other | 3.0
  Colostomy, temporary (n=32) | 47.50
  Colostomy, definitive (n=32) | 32.50
  No colostomy | 20.0

4. Secondary Outcome: Percentage of Participants With Complete Response (CR) at the End of Neoadjuvant Treatment
Description: Percentage of participants with CR was evaluated as the proportion of participants with complete response for the target and non-target lesions, separately, at the end of NAT according to the Response Evaluation Criteria in Solid Tumors (RECIST). CR was defined as disappearance of all target lesions or all non-target lesions and normalization of tumor marker levels.
Time Frame: BL and within 6 weeks after the completion of study treatment
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Bv+Capecitabine/Bv+Leucovorin+5-FU
Number analyzed (Participants) | 43
percentage of participants
  CR of target lesion(s) | 11.63
  CR of non-target lesion(s) | 18.60

5. Secondary Outcome: Percentage of Participants With an Overall Response of CR at the End of Neoadjuvant Treatment
Description: Percentage of participants with an overall response of CR was evaluated as the proportion of participants with CR for the target and non-target lesions plus absence of new lesions at the end of NAT according to RECIST. CR was defined as disappearance of all target lesions, all non-target lesions, and normalization of tumor marker levels.
Time Frame: BL and within 6 weeks after the completion of study treatment
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Bv+Capecitabine/Bv+Leucovorin+5-FU
Number analyzed (Participants) | 43
percentage of participants | 9.30

6. Secondary Outcome: Percentage of Participants With New Lesions at the Primary Tumor Site at the End of Neoadjuvant Treatment
Description: The percentage of participants with new lesions located at the primary tumor site were evaluated at the end of NAT.
Time Frame: BL and within 6 weeks after the completion of study treatment
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Bv+Capecitabine/Bv+Leucovorin+5-FU
Number analyzed (Participants) | 43
percentage of participants | 4.65

7. Secondary Outcome: Percentage of Participants With Relapse During Follow-Up
Description: The percentage of participants with local and/or regional relapse during follow-up. New lesions located at rectum or at colon or at lymph node detected at the end of NAT were evaluated as local and/or regional relapse.
Time Frame: BL, within 6 weeks after the completion of neoadjuvant treatment, every 2 weeks for 1 year following surgery, every 3 months thereafter until progression, up to 45 months
Population: ITT population; only participants who underwent radical surgery were included in the analysis
Measure: Number; unit: percentage of participants
Arm/Group | Bv+Capecitabine/Bv+Leucovorin+5-FU
Number analyzed (Participants) | 38
percentage of participants
  No Relapse | 84.21
  1 Relapse | 7.89
  2 Relapses | 7.89

8. Secondary Outcome: Disease-Free Survival (DFS) - Percentage of Participants With an Event
Description: DFS was defined as the time from treatment start date to the date of first progression of disease or date of death due to any cause.
Time Frame: as for outcome 7
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Bv+Capecitabine/Bv+Leucovorin+5-FU
Number analyzed (Participants) | 43
percentage of participants | 30.23

9. Secondary Outcome: DFS - Time to Event
Description: The time in months from date of start-of-treatment to the date of event defined as the first documented disease progression or death due to any cause. If a participant did not have an event, the time was censored at the date of last adequate tumor assessment. DFS was estimated using the Kaplan-Meier method.
Time Frame: as for outcome 7
Population: ITT population
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Bv+Capecitabine/Bv+Leucovorin+5-FU
Number analyzed (Participants) | 43
months | 27.43 (1.71)

10. Secondary Outcome: Overall Survival (OS) - Percentage of Participants With an Event
Description: OS was defined as the time from the date of first day of treatment until death due to any cause or the last date the participant was known to be alive.
Time Frame: BL, within 6 weeks after the completion of neoadjuvant treatment, every 2 weeks for 1 year following surgery, every 3 months thereafter until death, up to 45 months
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Bv+Capecitabine/Bv+Leucovorin+5-FU
Number analyzed (Participants) | 43
percentage of participants | 25.58

11. Secondary Outcome: OS - Time to Event
Description: OS was defined as the time from the date of first day of treatment until death due to any cause or the last date the participant was known to be alive. OS was estimated using the Kaplan-Meier method.
Time Frame: as for outcome 10
Population: ITT population
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Bv+Capecitabine/Bv+Leucovorin+5-FU
Number analyzed (Participants) | 43
months | 32.14 (1.46)

12. Secondary Outcome: Time to Disease Progression (TTP) - Percentage of Participants With an Event
Description: TTP was defined as the time from date of treatment start until first documented progression of disease or death due to underlying cancer.
Time Frame: as for outcome 10
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Bv+Capecitabine/Bv+Leucovorin+5-FU
Number analyzed (Participants) | 43
percentage of participants | 27.91

13. Secondary Outcome: TTP - Time to Event
Description: TTP was defined as the time from date of treatment start until first documented progression of disease or death due to underlying cancer. TTP was estimated using the Kaplan-Meier method.
Time Frame: as for outcome 10
Population: ITT population
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Bv+Capecitabine/Bv+Leucovorin+5-FU
Number analyzed (Participants) | 43
months | 27.68 (1.72)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the date of first study-drug administration until 28 days after the last dose of study drug administration.
Description: All enrolled participants who received at least 1 dose of study medication were included in the safety population.
Arm/Group | Bv+Capecitabine/Bv+Leucovorin+5-FU
Serious Adverse Events (participants affected / at risk) | 8/42
Other Adverse Events (participants affected / at risk) | 39/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bv+Capecitabine/Bv+Leucovorin+5-FU (N=42)
Diarrhoea (Gastrointestinal disorders) | 1
Miocardic ischemia (Cardiac disorders) | 1
Bowel perforation (Gastrointestinal disorders) | 1
Cardiac ischemia (Cardiac disorders) | 1
Anastomosis dehiscence (Injury, poisoning and procedural complications) | 1
Intestinal occlusion (Gastrointestinal disorders) | 1
Postoperative abscess (Injury, poisoning and procedural complications) | 1
Ipokaliemia (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bv+Capecitabine/Bv+Leucovorin+5-FU (N=42)
Anemia (Blood and lymphatic system disorders) | 5
Leukopenia (Blood and lymphatic system disorders) | 7
Neutropenia (Blood and lymphatic system disorders) | 6
Abdominal pain (Gastrointestinal disorders) | 6
Constipation (Gastrointestinal disorders) | 4
Diarrhea (Gastrointestinal disorders) | 18
Hematochezia (Gastrointestinal disorders) | 8
Nausea (Gastrointestinal disorders) | 9
Proctalgia (Gastrointestinal disorders) | 10
Proctitis (Gastrointestinal disorders) | 5
Rectal hemorrhage (Gastrointestinal disorders) | 3
Rectal tenesmus (Gastrointestinal disorders) | 7
Asthenia (General disorders) | 6
Fatigue (General disorders) | 4
Pyrexia (General disorders) | 3
Cystitis (Infections and infestations) | 4
Hypokalaemia (Metabolism and nutrition disorders) | 2
Dysuria (Renal and urinary disorders) | 3
Hypertension (Vascular disorders) | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Tachycardia (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 2
Conjunctivitis (Eye disorders) | 1
Anal fistula (Gastrointestinal disorders) | 1
Anorectal discomfort (Gastrointestinal disorders) | 2
Haemorrhoids (Gastrointestinal disorders) | 1
Mucous stools (Gastrointestinal disorders) | 2
Perianal erythema (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 2
Mucosal inflammation (General disorders) | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 2
Hypertransaminasaemia (Hepatobiliary disorders) | 1
Iatrogenic infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 1
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1
Blood lactate dehydrogenase increased (Investigations) | 1
Transaminases abnormal (Investigations) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Fistula (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 2
Neurotoxicity (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Strangury (Renal and urinary disorders) | 2
Prostatitis (Reproductive system and breast disorders) | 1
Vulvovaginal burning sensation (Reproductive system and breast disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal swelling (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Arterial thrombosis (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request the Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.